CLINICAL TRIAL: NCT07181681
Title: A Phase 1a/b Study to Investigate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Preliminary Antitumor Activity of BG-C0902, an Antibody-Drug Conjugate Targeting Epidermal Growth Factor Receptor (EGFR) × Mesenchymal-Epithelial Transition (MET), Alone and in Combination With Other Therapeutic Agents in Patients With Advanced Solid Tumors
Brief Title: A First-in-Human Study of BG-C0902 Alone and in Combination With Other Therapeutic Agents in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: BeOne Medicines (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BG-C0902-101
Record Dates: First submitted 2025-09-12; First posted 2025-09-18 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Solid Tumors; Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1a: Dose Escalation and Safety Expansion of BG-C0902 (Experimental): Sequential cohorts of increasing dose levels of BG-C0902 will be evaluated as monotherapy.
  Interventions: Drug: BG-C0902
- Phase 1b: Dose Expansion of BG-C0902 (Experimental): The recommended dose(s) for expansion (RDFE) for BG-C0902 from Part 1 will be evaluated in selected tumors.
  Interventions: Drug: BG-C0902

INTERVENTIONS:
Drug: BG-C0902 — Administered by intravenous infusion

SUMMARY:
This study is a first-in-human (FIH), Phase 1a/1b study of BG-C0902, a fully humanized anti-epidermal growth factor receptor (EGFR) and anti-mesenchymal-epithelial transition (MET) antibody, conjugated via an enzymatically cleavable linker to a topoisomerase 1 (TOPO1) inhibitor payload. The study aims to assess the safety, tolerability, pharmacokinetics (PK), pharmacodynamics, and preliminary antitumor activity of BG-C0902 in participants with advanced solid tumors. The study will be conducted in 2 phases: Phase 1a (dose escalation and safety expansion) and Phase 1b (dose expansion).

DETAILED DESCRIPTION:
Our company, previously known as BeiGene, is now officially BeOne Medicines. Because some of our older studies were sponsored under the name BeiGene, you may see both names used for this study on this website.

ELIGIBILITY:
Inclusion Criteria:

* Participants with histologically or cytologically confirmed advanced, metastatic, or unresectable solid tumors not amenable to therapy with curative intent or for whom treatment is not available or not tolerated.
* Participants must be able to provide archival tissue formalin-fixed paraffin-embedded (FFPE) block containing tumor tissue or approximately 10 to 15 freshly cut unstained FFPE slides) or recently obtained fresh tumor biopsy samples at screening.
* Participants must have ≥ 1 measurable lesion as assessed by RECIST v1.1.
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 1, as assessed ≤ 14 days before the first dose of study drug.
* Adequate bone marrow and organ function as indicated by the following laboratory values ≤ 14 days before the first dose of study drug
* Female participants of childbearing potential must be willing to use a highly effective method of birth control for the duration of the study and for ≥ 7 months after the last dose of study drug. They must also have a negative serum pregnancy test result ≤ 3 days before the first dose of study drug.
* Nonsterile male participants must be willing to use a highly effective method of birth control and refrain from sperm donation for the duration of the study and for ≥ 4 months after the last dose of study drug.

Exclusion Criteria:

* History of severe allergic reactions or hypersensitivity to BG-T187 or other monoclonal antibodies, or to the active ingredient and excipients of the study drug or camptothecins.
* For Phase 1a Part B Safety Expansion and Phase 1b only: Prior treatment with an EGFR-targeting ADC or mesenchymal-epithelial transition (MET)-targeting antibody-drug conjugate (ADC), or any ADC with topoisomerase I (TOPO1) inhibitor payload.
* Active leptomeningeal disease or uncontrolled, untreated brain metastasis. Participants with a history of treated and, at the time of screening, stable central nervous system (CNS) metastases are eligible, provided they meet all the following:

  1. Brain imaging at screening shows no evidence of interim progression, is clinically stable for ≥ 4 weeks, and has no evidence of new brain metastases
  2. Have measurable disease and/or evaluable disease outside CNS
  3. No ongoing requirement for corticosteroids as therapy for CNS disease; off corticosteroids ≥ 14 days before dosing with study drug; anticonvulsants at a stable dose are allowed
  4. No stereotactic radiation or whole-brain radiation ≤ 14 days before the first dose of study drug
* History of interstitial lung disease (ILD), or ≥ Grade 2 noninfectious pneumonitis ≤ 2 years before the first dose of the study drug, or has current ILD/noninfectious pneumonitis, or where suspected active ILD/noninfectious pneumonitis cannot be ruled out by imaging during screening.
* Participants with active or chronic corneal disorder, including but not limited to Sjögren's, Fuch's corneal dystrophy, history of corneal transplantation, corneal keratitis, keratoconjunctivitis, keratopathy, corneal abrasion, inflammation or ulceration, other active ocular conditions and any clinically significant corneal disease that prevents adequate monitoring of drug-induced keratopathy.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2025-11-10 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Phase 1a: Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Approximately 24 Months
Phase 1a: Number of Participants with Dose Limiting Toxicities (DLTs) | Approximately 21 Days
Phase 1a: Maximum Tolerated Dose (MTD) or Maximum Administered Dose (MAD) of BG-C0902 | Approximately 24 Months
  MTD is defined as the highest dose evaluated for which estimated toxicity rate is the closest to the target toxicity rate. MAD is defined as the highest dose administered if MTD is not reached.
Phase 1a: Recommended dose(s) for Expansion (RDFE) of BG-C0902 | Approximately 24 Months
  RDFE of BG-C0902 will be determined based upon the MTD or MAD.
Phase 1b: Recommended Phase 2 Dose (RP2D) of BG-C0902 as Monotherapy | Approximately 24 Months
  RP2D as determined based on safety, pharmacokinetics (PK), pharmacodynamics, preliminary antitumor activity, and other relevant data, as available.
Phase 1b: Overall Response Rate (ORR) | Approximately 24 Months
  ORR is defined as the percentage of participants with best overall response of complete response (CR) or partial response (PR) as determined from tumor assessments by the investigator using Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.

SECONDARY OUTCOMES:
Phase 1a: ORR | Approximately 24 Months
  ORR is defined as the percentage of participants with best overall response of CR or PR. as assessed by the investigator using RECIST v1.1.
Phase 1a and 1b: Duration of Response (DOR) | Approximately 24 Months
  DOR is defined as the time from the first confirmed objective response by the investigator using RECIST v1.1 until the first documentation of disease progression after treatment initiation or death, whichever comes first.
Phase 1a and 1b: Disease Control Rate (DCR) | Approximately 24 Months
  DCR is defined as the percentage of participants with the best overall response, of a CR, PR, and stable disease assessed by the investigator using RECIST v1.1.
Phase 1b: Progression-free Survival (PFS) | Approximately 24 Months
  PFS is defined as the time from first dose until first documentation of progression or death, whichever comes first, as assessed by the investigator using RECIST v1.1
Phase 1b: Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Approximately 24 Months
  Number of participants with treatment-emergent AEs and SAEs.
Phase 1a and 1b: Area under the Concentration-time Curve (AUC) of BG-C0902, Total Antibody, and Payload | Two times in the first three months
Phase 1a and 1b: Maximum Observed Plasma Concentration (Cmax) of BG-C0902, Total Antibody, and Payload | Two times in the first three months
Phase 1a and 1b: Time to Maximum Concentration (Tmax) of BG-C0902, Total Antibody, and Payload | Two times in the first three months
Phase 1a and 1b: Half-life (t1/2) of BG-C0902, Total Antibody, and Payload | Two times in the first three months
Phase 1a and 1b: Volume of Distribution (Vd) of BG-C0902, Total Antibody, and Payload | Two times in the first three months
Phase 1a and 1b: Number of Participants with Anti-drug Antibodies (ADAs) to BG-C0902 | Approximately 24 Months

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeOne Medicines
Locations (4):
- Next Oncology, Austin, Texas, United States
- Australia (2):
  - Blacktown Cancer and Haematology Centre, Blacktown, New South Wales
  - The Alfred Hospital, Melbourne, Victoria
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
BeOne shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe. Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved.
  BeOne shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations.
  Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for BeOne review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://beonemedicines.com/science/clinical-trials/